CLINICAL TRIAL: NCT05072158
Title: Pelvic Floor Disorders Among Sexual Minoritized Women
Acronym: PRIDE
Status: Terminated | Type: Observational
Why Stopped: PI has confirmed this is not a clinical trial and was entered in error in the system.
Sponsor: University of New Mexico (Other)
Collaborators: Albany Medical College (Other); University of Texas at Austin (Other)
Responsible Party: Sponsor
Other Study IDs: 21-196
Record Dates: First submitted 2021-08-18; First posted 2021-10-08 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Sexual Function Disturbances; Pelvic Organ Prolapse; Urinary Incontinence; Fecal Incontinence
MeSH Terms: conditions — Sexual Dysfunctions, Psychological; Pelvic Organ Prolapse; Urinary Incontinence; Fecal Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: None, this is an observational study — This is a qualitative study, we will be asking for patient experiences with PFDs and the impact on their sexual function.

SUMMARY:
The investigators aim to perform cognitive interviews to assess how pelvic floor disorders impact sexual functioning in women who have sex with women (WSW). As a secondary objective there will be cognitive interviews to assess perceptions of sexual function questionnaires such as Female Sexual Function Index (FSFI) and Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire-IUGA Revised (PISQ-IR) in WSW.

DETAILED DESCRIPTION:
There is a paucity of data regarding care of women who have sex with women (WSW). While some cohort studies are being performed in general gynecology, no studies document the reasons as to why WSW seek urogynecological care, or how pelvic floor disorders (PFDs) affect sexual function in this population. Another detrimental gap in current knowledge and a barrier to care for WSW is the lack of understanding of what would drive WSW to seek care, if there are special considerations for care, or if the commonly used condition specific questionnaires adequately reflect their concerns. The Investigators aim to perform qualitative interviews to understand how PFDs affect sexual function, and if commonly utilized sexual function questionnaires are inclusive to WSW.

ELIGIBILITY:
Inclusion Criteria:

* WSW who have a PFD (pelvic organ prolapse, urinary incontinence, fecal incontinence)
* Age >18
* Able to provide consent
* Able to read/write in English

Exclusion Criteria:

* WSW who have not been sexually active in the past 6 months
* Incarcerated patients
* Pregnant or lactating patients
* Unable to consent with study procedures or guided discussions
* Unable to speak English
* No sexual activity in the past 6 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This trial is open only to wmen
Study Population: New patients over the age of 18 who present to urogynecology office or contact the research team with interest in participating in the study who self-identify as women who have sex with women. This may include but is not limited to: lesbian and bisexual women.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2022-06-29 (Actual); Study Completion 2022-06-29 (Actual)

PRIMARY OUTCOMES:
Qualitative impact of pelvic floor disorders on sexual function | 6 months
  We will assess the impact of pelvic floor disorders with qualitative analysis and informational interviews

SECONDARY OUTCOMES:
Qualitative inclusivity of sexual function questionnaires | 6 months
  We will examine this with guided focus groups

CONTACTS AND LOCATIONS:
Overall Officials: Sierra Jansen, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No